CLINICAL TRIAL: NCT05464511
Title: Impact of Steerable Delivery Sheaths on Successful Closure of Left Atrial Appendage With AMULET Dual Mechanism Closure Device (STEER-CLOSE Study)
Brief Title: Impact of Steerable Delivery Sheaths on Successful Closure of LA A With AMULET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Collaborators: Kansas City Heart Rhythm Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCHRRF-STEERRCLOSE-0015
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Intervention Model Description: This will be a multi-centered, retrospective as well as prospective observational registry with patients undergoing LAAO with the dual mechanism closure Amulet device. This study will proceed with a target of 300 patients who have undergone or are planned to undergo LAAO with dual mechanism closure Amulet device. Patient level data of participating centers will be obtained from National Cardiovascular Data Registry (NCDR®) of patients who have already had the procedure. Prospective data will be collected for all patients willing to participate in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Amulet device using non-steerable fixed curve sheath (No Intervention): Patients undergoing left atrial appendage occlusion with the dual mechanism closure Amulet device using non-steerable fixed curve sheath.
- Patients with Amulet device using a novel steerable sheath (Active Comparator): Patients undergoing left atrial appendage occlusion with the dual mechanism closure Amulet device using a novel steerable sheath.
  Interventions: Other: Left atrial appendage occlusion with the dual mechanism closure Amulet device using a novel steerable sheath.

INTERVENTIONS:
Other: Left atrial appendage occlusion with the dual mechanism closure Amulet device using a novel steerable sheath. — Left atrial appendage occlusion with the dual mechanism closure Amulet device using a novel steerable sheath.
  Arms: Patients with Amulet device using a novel steerable sheath

SUMMARY:
The novel Amplatzer steerable delivery sheath (Abbott Vascular) is found to be safe and effective in performing LAAO procedure. However, the procedural outcomes have not been compared with the traditional non-steerable fixed curve sheath. In this study investigators aim to compare the outcome of patients undergoing left atrial appendage occlusion with the dual mechanism closure Amulet device using non-steerable fixed curve sheath versus a novel steerable sheath.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common abnormal heart rhythm associated with substantial morbidity and mortality. It is one of the strongest risk factors of systemic thromboembolism (TE), with stroke being the most serious outcome. Prevention of stroke is the cornerstone of managing AF, which can be achieved either by oral anticoagulation (OAC) or Percutaneous left atrial appendage occlusion (LAAO) in patients who have a contraindication to OAC. Heterogeneity in cardiac chamber size, interatrial septum, LAA anatomy and orientation, operator experience and currently available fixed curve sheaths add to the complexity of the procedure. Alignment of LAAO device along the access of the left atrial appendage body is an important factor in improving closure rates. The devices which are currently approved by FDA for LAA closure in the U.S. are Amplatzer Amulet device (Abbott Medical) and Watchman and Watchman FLX devices (Boston Scientific). In a recent study, Amplatzer Amulet device was found to be noninferior in terms of safety and effectiveness, with superior LAA occlusion rates but higher device-related complications as compared to first generation watchman device. The LAAO device sheaths that are used currently have fixed shapes and angles that may not be optimal for some LAA anatomy, which can lead to excessive device manipulation, prolonged procedure time, and potentially suboptimal co-axiality during the process. This may lead to increase device related complications. The new Amplatzer steerable delivery sheath (Abbott Vascular) is designed to provide distal bidirectional steerability of the sheath for Amulet implantation. Such steerability may enable successful endovascular closure of greater proportion of LAA, allow precise position of the transseptal puncture, and potentially reduce procedural times and complications with complex cases.

Investigators hypothesize that the use of novel steerable sheath for LAAO closure is safer and more effective as compared to non-steerable fixed curve sheath

ELIGIBILITY:
Inclusion Criteria:

Patients with atrial fibrillation who meets the indication/criteria for left atrial appendage occlusion and undergoing implantation of Amplatzer™ Amulet™ Left Atrial Appendage Occluder device

Exclusion Criteria:

* Patient been/being implanted with device other than Amplatzer™ Amulet™ Left Atrial Appendage Occluder
* Pregnant or breastfeeding patients
* Prisoners
* Patients not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Acute Closure of Left Atrial Appendage | 1 day
  Acute closure ( less than or equal to 3mm) of the left atrial appendage after Left Atrial Appedage Occlusion(LAAO) procedure
Number of patients with Cardiac Perforation | 7 days
  Number of patients with cardiac perforation
Need for Pericardiocentesis | 7 days
  Need for pericardiocentesis within 7 days of implantation

SECONDARY OUTCOMES:
Number of devices | 1 day (procedure day)
  Number of devices changed prior to final implant during the procedure
Number of device repositions | 1 day (procedure day)
  Number of device repositions performed during the procedure
Closure Rates | 45 days
  45 day closure rates of left atrial appendage ( less than or equal to 3mm)
Number of participants with Device related thrombus (DRT) | 45 days
  Number of participants with Device related thrombus (DRT)
Number of participants with Transient ischemic attack (TIA) or cerebrovascular accident (CVA) | 6 months
  Number of participants with Transient ischemic attack (TIA) or cerebrovascular accident (CVA) within 6 months of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (7):
- United States (7):
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas
  - Centerpoint Medical Center Clinic, Independence, Missouri
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center Clinic, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gangireddy SR, Halperin JL, Fuster V, Reddy VY. Percutaneous left atrial appendage closure for stroke prevention in patients with atrial fibrillation: an assessment of net clinical benefit. Eur Heart J. 2012 Nov;33(21):2700-8. doi: 10.1093/eurheartj/ehs292. Epub 2012 Sep 24. PMID 23008509
- [Background] Reddy VY, Sievert H, Halperin J, Doshi SK, Buchbinder M, Neuzil P, Huber K, Whisenant B, Kar S, Swarup V, Gordon N, Holmes D; PROTECT AF Steering Committee and Investigators. Percutaneous left atrial appendage closure vs warfarin for atrial fibrillation: a randomized clinical trial. JAMA. 2014 Nov 19;312(19):1988-98. doi: 10.1001/jama.2014.15192. PMID 25399274
- [Background] Jazayeri MA, Vuddanda V, Parikh V, Lakkireddy DR. Percutaneous left atrial appendage closure: current state of the art. Curr Opin Cardiol. 2017 Jan;32(1):27-38. doi: 10.1097/HCO.0000000000000367. PMID 27898435
- [Background] Lakkireddy D, Thaler D, Ellis CR, Swarup V, Sondergaard L, Carroll J, Gold MR, Hermiller J, Diener HC, Schmidt B, MacDonald L, Mansour M, Maini B, O'Brien L, Windecker S. Amplatzer Amulet Left Atrial Appendage Occluder Versus Watchman Device for Stroke Prophylaxis (Amulet IDE): A Randomized, Controlled Trial. Circulation. 2021 Nov 9;144(19):1543-1552. doi: 10.1161/CIRCULATIONAHA.121.057063. Epub 2021 Aug 30. PMID 34459659
- [Background] Saw J, Perrin N, Nestelberger T, Mondesert B, Tsang M, Ibrahim R. First-in-Human Experience With the Amplatzer Steerable Delivery Sheath for Left Atrial Appendage Closure. JACC Cardiovasc Interv. 2021 Oct 11;14(19):2191-2193. doi: 10.1016/j.jcin.2021.07.022. No abstract available. PMID 34620400